CLINICAL TRIAL: NCT01445535
Title: Phase 1 Trial of Siplizumab and Dose-Adjusted EPOCH-Rituximab (DA-EPOCH-R) in T and NK-Cell Lymphomas
Brief Title: Phase 1 Trial of Siplizumab and Dose-Adjusted EPOCH-Rituximab in T- and NK-Cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wyndham Wilson, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 090065; 09-C-0065; NCT00832936 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: T-Cell Peripheral Lymphoma; Gamma Delta Hepatosplenic T-Cell Lymphoma; Subcutaneous Panniculitis-Like T-Cell Lymphoma; NK T-Cell Lymphoma
Keywords: CD2 Positive; Toxicity; EBV Lymphoma; Chemotherapy Naive; Maximum Tolerated Dose; Lymphoma; T-Cell Lymphoma; NK T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Subcutaneous panniculitis-like T-cell lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma; Lymphoma, T-Cell | interventions — Rituximab; Etoposide; siplizumab; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- siplizumab + EPOCH (combo chemo) + rituximab (Experimental): siplizumab will be given with EPOCH (combo chemo) and rituximab every 21 days
  Interventions: Biological: Rituximab; Drug: Etoposide; Biological: Siplizumab; Drug: Prednisone; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Doxorubicin

INTERVENTIONS:
Biological: Rituximab — Rituximab will be given with siplizumab and etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin every 21 days
  Other Names: Rituxan
Drug: Etoposide — Etoposide will be given with siplizumab and prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab every 21 days
  Other Names: Toposar
Biological: Siplizumab — Siplizumab will be given with etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab every 21 days
  Other Names: MEDI-507
Drug: Prednisone — Prednisone will be given with siplizumab and etoposide, vincristine, cyclophosphamide, doxorubicin and rituximab every 21 days
  Other Names: Deltasone
Drug: Vincristine — Vincristine will be given with siplizumab and etoposide, prednisone, cyclophosphamide, doxorubicin and rituximab every 21 days
  Other Names: Marqibo
Drug: Cyclophosphamide — Cyclophosphamide will be given with siplizumab and etoposide, prednisone, vincristine, doxorubicin and rituximab every 21 days
  Other Names: Cytoxan
Drug: Doxorubicin — Doxorubicin will be given with siplizumab and etoposide, prednisone, cyclophosphamide and rituximab every 21 days
  Other Names: Doxil

SUMMARY:
Studies conducted at the National Cancer Institute suggest that certain chemotherapy drugs may be more effective if given by continuous infusion into the vein rather than by the standard method of rapid intravenous injection. One such combination of six chemotherapy drugs, known as Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, Rituximab (EPOCH-R), has had a high degree of effectiveness in people with certain kinds of cancer. Recent evidence also indicates that the effects of chemotherapy may be improved by combining the treatment with monoclonal antibodies, which are purified proteins that are specially made to attach to foreign substances such as cancer cells. This protocol is specifically for adults with the types of cancer known as T-cell and Naturel Killer (NK)-cell lymphomas, who have never received chemotherapy previously. The additional monoclonal antibody in the study, called siplizumab, has been manufactured to attach to the cluster of differentiation 2 (CD2) protein contained in these types of tumors.

Study volunteers will need to undergo an initial period of evaluation that may take up to 3 weeks and may be done on an outpatient basis. Evaluation may include some or all of the following tests: blood and urine tests, tests of lung and heart function, lumbar punctures to take samples of cerebrospinal fluid, magnetic resonance imaging (MRI) or computerized tomography (CT) scans, full-body positron emission tomography (PET) scans, bone marrow biopsies, and biopsies of suspected tumor areas.

During the study, patients will receive EPOCH-R chemotherapy, which includes the following drugs: etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab. The additional drug, siplizumab, will be given by IV infusion on the first day of treatment over several hours. When the siplizumab intravenous (IV) infusion is complete, the drugs doxorubicin, etoposide, and vincristine will each be given by continuous IV infusion over the next 4 days (that is, continuously for a total of 96 hours). When this infusion is completed, the drugs rituximab and cyclophosphamide will be given by IV infusion over several hours on Day 5. Prednisone will be given by mouth twice each day for 5 days. Patients may be given other drugs to treat the side effects of chemotherapy and to prevent possible infections.

The siplizumab-EPOCH-R therapy will be repeated every 21 days, which is known as a cycle of therapy, for a total of 6 cycles. Following the fourth and sixth treatment cycles (approximately weeks 12 and 18) of siplizumab-EPOCH-R, study researchers will perform blood tests and CT/MRI scans on all patients to assess their response to the treatment.

DETAILED DESCRIPTION:
Background:

The clinical outcome for patients with T-cell non-Hodgkin's lymphoma is significantly inferior to the outcome of patients with B-cell non-Hodgkin's lymphoma. In most reports less than 20% of patients with T cell lymphoid malignancies remain free of disease at 5 years.

The combination of alemtuzumab and Etoposide, Prednisone, Vincristine, Cyclophosphamide and Doxorubicin (EPOCH) chemotherapy was evaluated in patients with chemotherapy naive aggressive T and natural killer (NK) cell lymphoid malignancy. Dose-limiting bone marrow toxicity prevented escalation of the alemtuzumab dose.

Siplizumab is a humanized monoclonal antibody directed at cluster of differentiation 2 (CD2) that demonstrated activity in the treatment of relapsed/refractory T cell lymphoma, suggesting further development by combining with chemotherapy for untreated patients. Siplizumab caused Epstein-Barr Virus (EBV) lymphoproliferative disease in patients treated with a weekly schedule of administration.

Rituximab prevents the development of EBV lymphoproliferative disease in the allogeneic transplant setting and may be active in preventing EBV-related B cell lymphoma in other settings.

Objectives:

Determine the toxicity and maximum tolerated dose of siplizumab and dose-adjusted EPOCH rituximab chemotherapy in chemotherapy naïve CD2- expressing T and NK lymphoid malignancies.

Eligibility:

CD2-expressing lymphoid malignancy.

Patients with chemotherapy naive aggressive T & NK lymphomas. Patients with alk-positive anaplastic large cell lymphoma and patients with T-cell precursor disease are not eligible.

Design:

Four dose levels of siplizumab will be evaluated to determine the toxicity profile and in a preliminary fashion, and its activity in combination with dose-adjusted EPOCH with rituximab.

Four dose levels of siplizumab will be explored, in cohorts of three to six patients each. Patients will receive 3.4, 4.8, 8.5, or 15 mg/kg of siplizumab on day 1 of therapy, followed by dose-adjusted EPOCH-rituximab chemotherapy days 1-5 every 3 weeks for a total of 6 cycles.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cluster of differentiation 2 (CD2)-expressing lymphoid malignancy, confirmed by pathology or flow cytometry staff of the Hematopathology Section, Laboratory of Pathology, National Cancer Institute (NCI). At least 30% of the malignant cells must be CD2 positive for inclusion in this study.

Patients with chemotherapy naive T & Natural Killer (NK) lymphomas, including but not limited to peripheral T cell lymphoma (nos), gamma-delta hepatosplenic T cell lymphoma, subcutaneous panniculitis-like T cell, NK-T cell lymphoma confirmed by pathology or flow cytometry staff of the Hematopathology Section, Laboratory of Pathology, NCI. Patients with alk-positive anaplastic large cell lymphoma and patients with T-cell precursor disease are not eligible.

Age greater than or equal to 18 years.

Laboratory tests: Creatinine less than or equal to 1.5 mg/dL or creatinine clearance greater than or equal to 60 ml/min; bilirubin less than 2.0 mg/dl unless due to Gilbert's (unconjugated hyperbilirubinemia without other known cause), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 times upper limit of normal (ULN) (AST and ALT less than or equal to 6 times ULN for patients on hyperalimentation for whom these abnormalities are felt to be due to the hyperalimentation) and; Absolute neutrophil count (ANC) greater than or equal to 1000/mm(3), platelet greater than or equal to 75,000/mm(3); unless impairment due to respective organ impairment by tumor.

No active symptomatic ischemic heart disease, myocardial infarction or congestive heart failure within the past year.

Patients must not have a marked baseline prolongation of Q wave, T wave (QT/QTc) interval (e.g., demonstration of a corrected QT interval (QTc) interval >500 milliseconds (ms)).

Human immunodeficiency virus (HIV) negative, because of the unknown effects of combined therapy with chemotherapy and an immunosuppressive agent on HIV progression.

Signed informed consent by the patient or patient's representative.

Willing to use contraception.

Not pregnant or nursing, because of the unknown effects of dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R) or siplizumab on the developing fetus and infant.

No serious underlying medical condition or infection that would contraindicate treatment. Patients with central nervous system (CNS) involvement are eligible for treatment on this study.

EXCLUSION CRITERIA:

Patients less than 18 years of age will be excluded because siplizumab has not been given to minors in combination with chemotherapy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01-13 (Actual); Primary Completion 2011-04-01 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H Wilson, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abruzzo LV, Rosales CM, Medeiros LJ, Vega F, Luthra R, Manning JT, Keating MJ, Jones D. Epstein-Barr virus-positive B-cell lymphoproliferative disorders arising in immunodeficient patients previously treated with fludarabine for low-grade B-cell neoplasms. Am J Surg Pathol. 2002 May;26(5):630-6. doi: 10.1097/00000478-200205000-00009. PMID 11979093
- [Background] Bhargava R, Barbashina V, Filippa DA, Teruya-Feldstein J. Epstein-Barr virus positive large B-cell lymphoma arising in a patient previously treated with Cladribine for hairy cell leukemia. Leuk Lymphoma. 2004 May;45(5):1043-8. doi: 10.1080/10428190310001625890. PMID 15291365
- [Background] Birkeland SA, Hamilton-Dutoit S. Is posttransplant lymphoproliferative disorder (PTLD) caused by any specific immunosuppressive drug or by the transplantation per se? Transplantation. 2003 Sep 27;76(6):984-8. doi: 10.1097/01.TP.0000085602.22498.CF. PMID 14508366
- [Result] Roswarski J, Roschewski M, Lucas A, Melani C, Pittaluga S, Jaffe ES, Steinberg SM, Waldmann TA, Wilson WH. Phase I dose escalation study of the anti-CD2 monoclonal antibody, siplizumab, with DA-EPOCH-R in aggressive peripheral T-cell lymphomas. Leuk Lymphoma. 2018 Jun;59(6):1466-1469. doi: 10.1080/10428194.2017.1387908. Epub 2017 Oct 16. No abstract available. PMID 29032710
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0065.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - 3.4 mg/kg: 3.4 mg/kg siplizumab was given on day 1 of each cycle followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH) (combo chemo) on days 1-5 for 21 days.
- Cohort 2 - 4.8 mg/kg: 4.8 mg/kg siplizumab was given on day 1 of each cycle followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH) (combo chemo) on days 1-5 for 21 days.
- Cohort 3 - 8.5 mg/kg: 8.5 mg/kg siplizumab was given on day 1 of each cycle followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH) (combo chemo) on days 1-5 for 21 days.
- Cohort 4 - 15 mg/kg: 15 mg/kg siplizumab was given on day 1 of each cycle followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH) (combo chemo) on days 1-5 for 21 days.
Period: Overall Study
Arm/Group | Cohort 1 - 3.4 mg/kg | Cohort 2 - 4.8 mg/kg | Cohort 3 - 8.5 mg/kg | Cohort 4 - 15 mg/kg
Started | 3 | 3 | 3 | 6
Completed | 2 | 3 | 2 | 4
Not Completed | 1 | 0 | 1 | 2
Not completed — Enrolled/taken off study, no drug avail. | 0 | 0 | 0 | 1
Not completed — Disease progression | 1 | 0 | 1 | 0
Not completed — PI discretion | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 3.4 mg/kg | Cohort 2 - 4.8 mg/kg | Cohort 3 - 8.5 mg/kg | Cohort 4 - 15 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 0 | 4 | 10
  >=65 years | 0 | 0 | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.43 (16.1) | 42.2 (10.31) | 70.03 (6.87) | 45.38 (17.1) | 48.76 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 5 | 9
  Male | 0 | 3 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 4 | 4
  Not Hispanic or Latino | 3 | 3 | 3 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 2 | 8
  White | 1 | 1 | 1 | 4 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 6 | 15
Disease Status [Count of Participants; unit: Participants] — ATL: Adult T-cell leukemia/lymphoma; PTCL: peripheral T-cell lymphoma not-otherwise specified; EATL: enteropathy-associated T-cell lymphoma; CGDTCL: cutaneous gamma/delta T-cell lymphoma.
  Participants
    ATL | 2 | 1 | 2 | 3 | 8
    PTCL, NOS | 1 | 2 | 1 | 1 | 5
    EATL | 0 | 0 | 0 | 1 | 1
    CGDTCL | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed until 30 days after removal from study treatment or until off study, whichever comes first, approximately 22 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 3.4 mg/kg | Cohort 2 - 4.8 mg/kg | Cohort 3 - 8.5 mg/kg | Cohort 4 - 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 3 | 3 | 3 | 5

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Siplizumab
Description: A classic 3+3 dose-escalation design was used to assess the MTD of siplizumab in combination with dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R). If 2 of 6 patients experienced a dose-limiting toxicity (DLT) at a particular dose level, the MTD has been exceeded. The preceding dose level will be the MTD, provided 6 patients have been entered at this level and no more than one has experienced a DLT. DLTs for siplizumab was defined as infusional grade 3 non-hematologic toxicity lasting longer than 6 hours after the infusion, any grade 4 non-hematologic toxicity, or the development of an Epstein Barr Virus (EBV)-related lymphoproliferative disorder (LPD). Expected toxicities of dose-adjusted EPOCH-R and grade 3 laboratory adverse events (AEs) were not considered to be DLTs.
Time Frame: First 30 days after treatment initiation.
Measure: Number; unit: mg/kg
Groups:
- All Participants: All participants who received 3.4 mg/kg, 4.8 mg/kg, 8.5 mg/kg and 15 mg/kg siplizumab given on day 1 of each cycle followed by etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH) (combo chemo) on days 1-5 for 21 days.
Arm/Group | All Participants
Number analyzed (Participants) | 15
mg/kg | 15

3. Secondary Outcome: Number of Participants With a Response to Therapy
Description: Response was assessed by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma. Complete Remission was defined as the disappearance of all detectable clinical and radiographic evidence of disease, disappearance of all disease related symptoms if present before therapy, and normalization of those biochemical abnormalities (for example lactate dehydrogenase (LDH)) definitely assignable to the lymphoma. Complete response unconfirmed was defined as a residual node greater than 1.5 cm, with a decrease by greater than 75 percent in the sum of the products of the perpendicular diameters (SPD) of all measured lymph nodes. Partial Response was defined as a ≥ 50% decreased in SPD of 6 largest dominant nodes or nodal masses. Relapsed disease was defined as the appearance of any new lesion or increase by ≥50% in the size of the previously identified sites. Progressive disease was defined as a ≥50% increase from nadir in the SPD.
Time Frame: Response assessments were performed after the fourth and sixth cycle of therapy, at therapy completion, and every 3 months for year 1, four months for year 2, 6 months for years 3-5, and annually thereafter, up to 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 3.4 mg/kg | Cohort 2 - 4.8 mg/kg | Cohort 3 - 8.5 mg/kg | Cohort 4 - 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants
  Complete Remission | 1 | 2 | 1 | 4
  Complete Response Unconfirmed | 0 | 0 | 0 | 0
  Partial Response | 1 | 1 | 1 | 0
  Relapsed Disease | 0 | 0 | 0 | 0
  Progressive Disease | 1 | 0 | 1 | 0
  Stable Disease | 0 | 0 | 0 | 0
  Not Evaluable | 0 | 0 | 0 | 2

4. Secondary Outcome: Overall Progression Free Survival (PFS)
Description: Progression was assessed by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma. Progression is defined as ≥50% increase from nadir in the sum of the products of the perpendicular diameters (SPD) of any previously identified abnormal nodes for Partial Response's or non-responders. Progression-free survival (PFS) was determined from the on-study date until date of progression or last follow-up. The probability of PFS as a function of time was estimated by the Kaplan-Meier method.
Time Frame: On-study date until date of progression or last follow up, approximately 7 months.
Population: Data collected from participants receiving different dose levels were combined and analyzed as a single Arm/Group as pre-specified in the study protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 15
Months | 6.8 [2.9 to 27.1]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was determined from the on-study date until date of progression or last follow up. The probability of OS as a function of time was estimated by the Kaplan-Meier method.
Time Frame: On study date until date of death or last follow up, approximately 12 months.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 15
Months | 12.1 [6.7 to 30.7]

6. Other Pre Specified Outcome: Number of Dose-Limiting Toxicities (DLT)
Description: DLTs for siplizumab was defined as infusional grade 3 non-hematologic toxicity lasting longer than 6 hours after the infusion, any grade 4 non-hematologic toxicity, or the development of an EBV-related lymphoproliferative disorder (LPD). Expected toxicities of dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R) and grade 3 laboratory AEs were not considered to be DLTs.
Time Frame: First 30 days after treatment initiation.
Measure: Number; unit: Dose Limiting Toxicities
Arm/Group | Cohort 1 - 3.4 mg/kg | Cohort 2 - 4.8 mg/kg | Cohort 3 - 8.5 mg/kg | Cohort 4 - 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6
Dose Limiting Toxicities | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed until 30 days after removal from study treatment or until off study, whichever comes first, approximately 22 weeks.
Arm/Group | Cohort 1 - 3.4 mg/kg | Cohort 2 - 4.8 mg/kg | Cohort 3 - 8.5 mg/kg | Cohort 4 - 15 mg/kg
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/3 | 3/3 | 4/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 2/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 3.4 mg/kg (N=3) | Cohort 2 - 4.8 mg/kg (N=3) | Cohort 3 - 8.5 mg/kg (N=3) | Cohort 4 - 15 mg/kg (N=6)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 3.4 mg/kg (N=3) | Cohort 2 - 4.8 mg/kg (N=3) | Cohort 3 - 8.5 mg/kg (N=3) | Cohort 4 - 15 mg/kg (N=6)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (2) | 2 (2) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 2 (3) | 1 (1) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Febrile neutropenia (Infections and infestations) | 1 (1) | 1 (1) | 3 (5) | 3 (4) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3) | 1 (2) | 1 (3) | 4 (9)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Hemoglobin (Metabolism and nutrition disorders) | 3 (11) | 3 (18) | 3 (12) | 5 (20)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Insomnia (General disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Laryngeal nerve dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (14) | 3 (20) | 3 (12) | 5 (23)
Lymphopenia (Blood and lymphatic system disorders) | 3 (10) | 3 (16) | 3 (15) | 5 (22)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Mood alteration::Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 4 (6)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 2 (5) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 2 (3) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 3 (4) | 1 (1) | 3 (4) | 4 (5)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (13) | 3 (14) | 3 (10) | 5 (20)
Pain::Abdomen NOS (Gastrointestinal disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0)
Pain::Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2) | 0 (0) | 4 (6)
Pain::Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 4 (7)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain::Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain::Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 3 (11) | 3 (15) | 3 (10) | 5 (15)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GU::Urethra (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Dental/teeth/peridontal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Pain NOS (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (4) | 3 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 2 (3) | 1 (1)
Rigors/chills (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sweating (diaphoresis) (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
CD4 count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Cardiac troponin I (cTnI) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Catheter-related
Infection with normal ANC or Grade 1 or 2 neutrophils::Abdomen NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Middle ear (otitis media) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain::Lymph node (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain::Middle ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (9) | 2 (2)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GI::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — (ANC <1.0 x 10e9/L)::Blood
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular surface disease (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Chest wall (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain::Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash: dermatitis associated with radiation::Chemoradiation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (General disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT01445535/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT01445535/ICF_001.pdf